CLINICAL TRIAL: NCT03657056
Title: Focused Ultrasound Neuromodulation for Treatment of Temporal Lobe Epilepsy
Acronym: LIFUP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled and IRB record was closed
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Darin Dougherty, MD, Director, Division of Neurotherapeutics, Department of Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018P001352
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Low Intensity Ultrasound Pulsarions
Keywords: Epilepsy; Ultrasound
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from the normal population of patients being treated for temporal lobe epilepsy Massachusetts General Hospital.
  Patients identified as candidates for temporal lobe surgery by the clinical team will be notified via a letter that has been signed by a physician representative of the practice of their eligibility for the study. An administrator will follow-up on the letter with a phone call. The physician of potential participants will be notified of their eligibility for the study, and be provided with a copy of the consent form. A total of 3 participants will be enrolled in the project.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- BX Pulsar 1002 (Experimental): Low-Intensity Focused Ultrasound Pulsation (LIFUP) sonications will be conducted using the LIFUP experimental device BX Pulsar 1002 produced by the Brainsonix Corporation. For the purposes of safety LIFUP sonications will be initiated at the FDA limit for diagnostic ultrasound. However, the minimally effective dose in humans applications, according to (Lee et al., 2015), when derated is approximately 1125mW/cm2.
  Interventions: Device: BX Pulsar 1002

INTERVENTIONS:
Device: BX Pulsar 1002 — LIFUP will be administered to the temporal region on the side to undergo surgery, within the focus producing seizures. The ultrasound will be focused on the highest activity area within the temporal lobe. Functional MRI of the brain will be obtained throughout the LIFUP session.
  After the participant is fitted with the transducer they will be placed in the MRI machine and undergo a series of scans. After placing the transducer over the anterior tip of the temporal lobe the participant will undergo fMRI BOLD scans with LIFUP excitation (from (Lee et al., 2015): Tone Burst Duration = 2ms and Pulse Repetition Frequency = 250Hz) at four levels of intensity (720mW/cm2, 1440mW/cm2, 2880mW/cm2 and 5760mW/cm2). Before increasing the intensity, the transducer will be moved approximately 5mm posterior. After the last excitation scan the LIFUP parameters will be changed to inhibitory parameters (from (Yoo et al., 2011): Tone Burst Duration = 0.5ms and Pulse Repetition Frequency = 100Hz).
  Other Names: LIFUP

SUMMARY:
The aim of the proposed study is to assess the feasibility of using the BrainSonix BX Pulsar 1002 low-frequency and Low-Intensity Focused Ultrasound Pulsations (LIFUP) in human subjects suffering from intractable temporal lobe epilepsy. The patients selected will already be scheduled to undergo surgery for resection of the temporal lobe, and the investigational therapy will be applied to the temporal lobe at least one day prior to its scheduled removal. The study is intended to provide preliminary evidence of safety, and establish the feasibility of LIFUP treatment as evidenced by a modulation of the Blood-oxygenation level dependent (BOLD) signal in functional MRI (fMRI), and normal findings from histological examination of the resected brain tissue.

DETAILED DESCRIPTION:
Non-invasive and controllable suppression of regional brain activity may open new avenues for the treatment and management of epilepsy. There is good evidence that direct stimulation of epileptogenic sources can powerfully suppress seizure rates, but so far minimally invasive attempts have shown limited success. Currently, there are no approved non-invasive procedures for seizure suppression.

Focused ultrasound (FUS) is a promising new potential treatment, because it can target any region in the brain, regardless of depth, with high spatial specificity. FUS allows for the non-invasive delivery of acoustic energy to a well-localized and circumscribed brain region of a few millimeters in diameter, depositing mechanical or thermal energy. The possibility of transcranial application of FUS into deep brain areas has already been demonstrated by the strategic placement and operation of an array of multiple ultrasound transducers.

The ultrasound based BrainSonix device is a highly novel non-invasive alternative to direct stimulation. Capitalizing on non-invasive high-intensity focused ultrasound (HIFU), BrainSonix, using an animal model, found early evidence of selective suppression of regional neural activity in the brain. Importantly these effects were non-thermal and reversible. Further study is required to validate and characterize the degree of suppressive effects on epilepsy to ensure safe application in human subjects. Low Intensity Focused Ultrasound Pulsation (LIFUP) differs from HIFU because the intensities of ultrasound used are an order of magnitude lower than HIFU. Also, whereas ablative HIFU is administered continuously, LIFUP is administered in short pulses, which reduces energy deposition. The investigators' and others data have demonstrated that administration of ultrasound, as LIFUP, causes a significant, but reversible, neuromodulatory effect, while preventing the tissue from being thermally damaged.

Study Procedures

Visit 1 Assessment The initial assessment will be performed shortly after signing the consent form. The patient will meet with the clinician and baseline demographic information and general physical information will be collected. The patient will also undergo a psychiatric/neurological evaluation, including a neurological exam, and several neuropsychiatric questionnaires using the Brief Symptom Inventory (BSI) self-report, the Beck Depression Inventory (BDI) self-report, a neuropsychiatric battery of tests described in section 9.2.4 below, the Mini-International Neuropsychiatric Interview (MINI) and the Mini-Mental Status Assessment (MMSE). They will also be required to complete an Magnetic Resonance Imaging (MRI) screening questionnaire to detect the presence of any devices that might present a safety risk.

Visit 2 Treatment and Assessment At visit 2, the location of the epileptic focus will be determined based on previously performed studies as part of the individual's routine epilepsy evaluation. The location of the epileptic focus will be determined based on previously performed studies as part of the individual's routine epilepsy evaluation. Brain MRI, interictal electroencephalogram (EEG), ictal EEG, interictal positron emission tomography (PET), ictal PET, interictal single-photon emission computerized tomography (SPECT), ictal SPECT, interictal magnetoencephalography (MEG), ictal MEG, and magnetic resonance (MR) spectroscopy data may be available and utilized to determine each participant's epileptogenic zone.

LIFUP will be administered to the temporal region on the side to undergo surgery, within the focus producing seizures (as determined by the comprehensive epilepsy evaluation). LIFUP session will take place during the 7 days prior to the operation. See Section 8.2.1 for more details regarding the LIFUP Sonication procedure.

The subject's heart rate and blood pressure will be monitored during the procedure. Routine electrode electroencephalography (EEG) will be recorded immediately before and after the LIFUP sonication session. Recording will last approximately 60 minutes.

The same neurological exam and neuropsychiatric questionnaires using the Brief Symptom Inventory (BSI) self-report, the Beck Depression Inventory (BDI) self-report, and the neuropsychiatric battery of tests described above will be performed at Visit 2, as well. Testing will last approximately 2 hours.

LIFUP Sonication Procedure

Low-Intensity Focused Ultrasound Pulsation (LIFUP) sonications will be conducted using the LIFUP experimental device BX Pulsar 1002 produced by the Brainsonix Corporation. LIFUP will be administered to the temporal region on the side to undergo surgery, within the focus producing seizures (as determined by the comprehensive epilepsy evaluation). In addition the functional magnet resonance imaging (fMRI) recording will be done during the LIFUP to determine the target area of activity and to navigate the focus of the transducer to that area. The ultrasound will be focused on the highest activity area within the temporal lobe. Functional MRI of the brain will be obtained throughout the LIFUP session. Initially LIFUP will be administered below the minimum effective dose determined in previous animal experiments. Up to 8 sonications will be administered during the LIFUP session. The total dose of LIFUP is not to exceed 2 min. The total time within the MRI machine will be up to 90 minutes.

After the participant is fitted with the transducer they will be placed in the MRI machine and undergo a series of scans. After placing the transducer over the anterior tip of the temporal lobe the participant will undergo fMRI BOLD scans with LIFUP excitation: Tone Burst Duration = 2ms and Pulse Repetition Frequency = 250Hz) at four levels of intensity (720mW/cm2, 1440mW/cm2, 2880mW/cm2 and 5760mW/cm2). Before increasing the intensity, the transducer will be moved approximately 5mm posterior. The excitation scans will be analyzed immediately for evidence of BOLD activation. After the last excitation scan the LIFUP parameters will be changed to inhibitory parameters: Tone Burst Duration = 0.5ms and Pulse Repetition Frequency = 100Hz).

Surgical Resection and Histology After surgical resection of the anterior temporal lobe, histology will be performed on the resected tissue to look for evidence of tissue injury not characteristic of temporal lobe epilepsy or previously identified on the routine brain MRI.

Three Month Follow-up At three months the epilepsy surgeon will assess the healing of the surgical wounds and will conduct a Structural MR. The results will be reported back to the investigator.

Six Month Follow-up At six months the epilepsy surgeon will carry out a neurogical exam, and several neuropsychiatric questionnaires using the Brief Symptom Inventory (BSI) self-report, the Beck Depression Inventory (BDI) self-report, a neuropsychiatric battery of tests described in section 9.2.4 below, the MINI, and the Mini Mental Status Assessment.

Neuropsychiatric Battery of Tests The following battery of neuropsychiatric tests will be performed on the study subjects at one of the participant's standard clinical visits, as part of their standard clinical care and at visit 2 following the LIFUP sonication procedure. This battery of tests has been designed to not interfere with their standard clinical care. The Visit 2 scores will be compared to the Visit 1 (Baseline) scores to assess neuropsychiatric changes as a result of the LIFUP procedure.

Seizure Account Participants will be instructed to maintain a daily log of all seizures from the date of consenting until the date of the operation.

Heart Rate and Blood Pressure Monitoring The patient will be affixed with a heart rate monitor. A periodic blood pressure check will be performed if the heart rate increases more than 30% during or immediately after sonication. The investigators' lab has the capacity to measure those parameters in MRI. If the patient's blood pressure has also increased more than 10% then they will be withdrawn from the study.

EEG Monitoring Routine electrode electroencephalography (EEG) recorded immediately before and after the LIFUP sonication session. Recording will last approximately 60 minutes.

A 30-minute awake EEG using scalp electrodes placed according to the International 10-20 System of electrode placement will be performed immediately before and immediately after the LIFUP treatment.

Interim Safety Analysis The data will be analyzed after the first subject in order to determine subsequent treatment paradigm in the next 2 subjects. After the first participant, histology data will also be analyzed by the investigator. If the participant shows histological damage in the a category (i.e. apoptosis, irreversible blood brain barrier (BBB) disruption, ischemia) at a given intensity then the investigators will continue with the next cohort of 2 participants, but the investigators will no longer use that intensity, or higher intensities. If more than one participant shows histological damage in the same category at the lowest intensity (720mW/cm2), then the study will be stopped.

Biostatistical Analysis

Statistical analyses will be performed using SAS® v9.3 or higher (SAS Institute, Cary NC, USA).

All statistical analyses of safety and performance measures will be descriptive in nature. Continuous variables will be summarized by a mean, standard deviation, minimum, median and maximum, and categorical variables by a count and percentage. Confidence intervals will be provided where relevant.

If multiple evaluations are taken in a single patient, statistics described below will be appropriately modified to accommodate the within patient correlation.

Demographic, medical and clinical history variables will be tabulated. Continuous variables will be summarized by a mean, standard deviation, minimum, median and maximum, and categorical variables by a count and percentage.

The numbers of patients who were enrolled and completed each visit of the study will be provided, as well as the reasons for all enrollment discontinuations, grouped by major reason (e.g., lost to follow-up, adverse event). A list of discontinued patients, protocol deviations, and patients excluded from the efficacy analysis will be provided as well.

Histological results in the resected tissue of the anterior temporal lobe will be presented.

Comparison of all neurological assessment scores at the pre-treatment visit and at the post-treatment visit will be presented.

Comparison of the number of epileptiform discharges and Epileptiform Discharge frequency (DF) during a 30-minute period before and a 30-minute period after LIFUP will be presented.

Change in BOLD signal during or after LIFUP sonication will be presented.

Subjects who do not have valid data for the efficacy measures will be treated as missing values. No imputation is planned.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18 to 60 years old.
* Subjects with clinical evidence from their diagnostic evaluations of unilateral hippocampal - dysfunction and epileptogenicity, confirmed via intracarotid amobarbital procedure (IAP) and neuropsychological testing.
* Subjects with seizures that have been refractory to treatment with at least three currently marketed antiepileptic drugs.
* Subjects currently taking antiepileptic medications.
* Subjects with at least 3 seizures/month based on seizure diary.
* Subjects with epilepsy who would clearly benefit from surgical intervention.
* Subjects who have been offered an anterior-mesial temporal lobe resection, performed en-bloc, as treatment for medication refractory epilepsy. This includes both dominant or non-dominant mesial temporal lobe focal epilepsy.

Exclusion Criteria:

* Subjects with a cognitive or psychiatric disorder that limits the ability to give informed consent or are unable to cooperate with the testing.
* Subjects with dementia, delirium and psychotic symptoms.
* Subjects with ferromagnetic materials in the head.
* Subjects with severe cardiac disease, increased intracranial pressure, or a transcutaneous electrical nerve stimulation (TENS) unit.
* Subjects who exhibit primary generalized seizures or pseudoseizures.
* Subjects who have seizures secondary to drugs, alcohol, metabolic illness or progressive degenerative disease.
* Subjects who have experienced status epilepticus during the 3-week period prior to the LIFUP procedure.
* Subjects (females) who are pregnant.
* Patients who have had electrodes implanted in the brain that were not explanted at least 6 weeks prior to the LIFUP procedure.
* Patients who have had electrodes implanted into the focal point of the temporal lobe that is proposed for the ultrasonic stimulation using LIFUP.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
FMRI - (Change in BOLD signal) | 6 Months
  Change in BOLD signal during or after LIFUP sonication

CONTACTS AND LOCATIONS:
Overall Officials: Darin Dougherty, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hynynen K, Jolesz FA. Demonstration of potential noninvasive ultrasound brain therapy through an intact skull. Ultrasound Med Biol. 1998 Feb;24(2):275-83. doi: 10.1016/s0301-5629(97)00269-x. PMID 9550186
- [Background] Gavrilov LR, Tsirulnikov EM, Davies IA. Application of focused ultrasound for the stimulation of neural structures. Ultrasound Med Biol. 1996;22(2):179-92. doi: 10.1016/0301-5629(96)83782-3. PMID 8735528
- [Background] Tyler WJ, Tufail Y, Finsterwald M, Tauchmann ML, Olson EJ, Majestic C. Remote excitation of neuronal circuits using low-intensity, low-frequency ultrasound. PLoS One. 2008;3(10):e3511. doi: 10.1371/journal.pone.0003511. Epub 2008 Oct 29. PMID 18958151
- [Background] Min BK, Bystritsky A, Jung KI, Fischer K, Zhang Y, Maeng LS, Park SI, Chung YA, Jolesz FA, Yoo SS. Focused ultrasound-mediated suppression of chemically-induced acute epileptic EEG activity. BMC Neurosci. 2011 Mar 6;12:23. doi: 10.1186/1471-2202-12-23. PMID 21375781
- [Background] Yoo SS, Kim H, Min BK, Franck E, Park S. Transcranial focused ultrasound to the thalamus alters anesthesia time in rats. Neuroreport. 2011 Oct 26;22(15):783-7. doi: 10.1097/WNR.0b013e32834b2957. PMID 21876461
- [Background] Deffieux T, Younan Y, Wattiez N, Tanter M, Pouget P, Aubry JF. Low-intensity focused ultrasound modulates monkey visuomotor behavior. Curr Biol. 2013 Dec 2;23(23):2430-3. doi: 10.1016/j.cub.2013.10.029. Epub 2013 Nov 14. PMID 24239121
- [Background] Lee W, Kim H, Jung Y, Song IU, Chung YA, Yoo SS. Image-guided transcranial focused ultrasound stimulates human primary somatosensory cortex. Sci Rep. 2015 Mar 4;5:8743. doi: 10.1038/srep08743. PMID 25735418
- [Background] Legon W, Sato TF, Opitz A, Mueller J, Barbour A, Williams A, Tyler WJ. Transcranial focused ultrasound modulates the activity of primary somatosensory cortex in humans. Nat Neurosci. 2014 Feb;17(2):322-9. doi: 10.1038/nn.3620. Epub 2014 Jan 12. PMID 24413698
- [Background] Mitchell LA, Jackson GD, Kalnins RM, Saling MM, Fitt GJ, Ashpole RD, Berkovic SF. Anterior temporal abnormality in temporal lobe epilepsy: a quantitative MRI and histopathologic study. Neurology. 1999 Jan 15;52(2):327-36. doi: 10.1212/wnl.52.2.327. PMID 9932952
- [Background] Vykhodtseva NI, Hynynen K, Damianou C. Histologic effects of high intensity pulsed ultrasound exposure with subharmonic emission in rabbit brain in vivo. Ultrasound Med Biol. 1995;21(7):969-79. doi: 10.1016/0301-5629(95)00038-s. PMID 7491751
- [Background] Vykhodtseva N, McDannold N, Martin H, Bronson RT, Hynynen K. Apoptosis in ultrasound-produced threshold lesions in the rabbit brain. Ultrasound Med Biol. 2001 Jan;27(1):111-7. doi: 10.1016/s0301-5629(00)00275-1. PMID 11295277
- [Background] Cohen MS, DuBois RM. Stability, repeatability, and the expression of signal magnitude in functional magnetic resonance imaging. J Magn Reson Imaging. 1999 Jul;10(1):33-40. doi: 10.1002/(sici)1522-2586(199907)10:13.0.co;2-n. PMID 10398975
- [Background] Smith SM, Jenkinson M, Woolrich MW, Beckmann CF, Behrens TE, Johansen-Berg H, Bannister PR, De Luca M, Drobnjak I, Flitney DE, Niazy RK, Saunders J, Vickers J, Zhang Y, De Stefano N, Brady JM, Matthews PM. Advances in functional and structural MR image analysis and implementation as FSL. Neuroimage. 2004;23 Suppl 1:S208-19. doi: 10.1016/j.neuroimage.2004.07.051. PMID 15501092